CLINICAL TRIAL: NCT07088328
Title: Effect of Pentoxyphylline in Nephroprotection Following Perinatal Asphyxia: Randomized Controlled Trial
Brief Title: Nephroprotection Following Perinatal Asphyxia: Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Farag, Assistant professor of Pediatrics, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0108348
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Neonatal Encephalopathy; Pentoxifylline Adverse Reaction
Keywords: preterm infants; nephroprotection
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pentoxifylline group (Active Comparator): They will be given pentoxifylline as reno-protective drug (trentoximal, Egypharma ; E.D.A Reg.No.: 25276/2007) was administered intravenously to Neonates with perinatal hypoxia at 5mg/kg/hr given over 6 h daily for 3 consecutive days
  Interventions: Drug: Pentoxifylline
- Control group (Placebo Comparator): They will not be given pentoxifylline as reno-protective drug
  Interventions: Other: placebo distilled water

INTERVENTIONS:
Drug: Pentoxifylline — Intravenous administration for 3 days
  Arms: Pentoxifylline group
Other: placebo distilled water — Intravenous administration for 3 days
  Arms: Control group

SUMMARY:
The aim of this study is to determine the value of Pentoxifylline for nephroprotection in these neonates with perinatal asphyxia, using cystatin C, regional oxygenation measured near infrared spectroscopy and renal Doppler sonography.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

1. Evidence of perinatal hypoxia, as indicated by at least one of the following:

   1. Apgar score of less than or equal to 5 at 10 minutes.
   2. ongoing resuscitation at 10 minutes.
   3. pH less than 7.14 or a base deficit worse than or equal to minus 12 mmol/L on cord/arterial/venous/capillary blood gas obtained within 60 minutes of birth.
2. Evidence of moderate to severe encephalopathy using Sarnat staging score.(14)
3. Greater than or equal to 35 weeks gestational age.
4. Birth weight greater than or equal to 1800 g.

Exclusion Criteria:

Neonates with any of the following will be excluded:

1. Birth weight less than 1800 g. 2. Major congenital malformations/chromosomal anomalies including major cardiac anomalies. 3. Preterm less than 35 weeks gestational age according to modified Ballard score. (15) 4. progressive neuromuscular disorders (eg spinal muscle atrophy). 5. Severe systemic infections (eg TORCH infection).

-

Ages: 1 Hour to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Renal function | daily in the first 3 days of life.
  creatinine level in mg/dl.

SECONDARY OUTCOMES:
Renal Doppler sonography | first 3 days of life
  Peak systolic velocity (PSV) in cm/sec End diastolic velocity (EDV) in cm/sec.
cystatin C | first 24 hours of life
  measure level using ng/L

IPD SHARING:
Plan to Share IPD: Undecided